CLINICAL TRIAL: NCT06535451
Title: Lung Cancer Early Detection With Low-dose Computed Tomography in High-risk Individuals: Experience in Mexico
Brief Title: Lung Cancer Screening Program in Mexico
Acronym: DETECTO
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Head of Thoracic Oncology Unit, Instituto Nacional de Cancerologia de Mexico
Other Study IDs: (015/005/ICI)(CEI 946/15)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
Keywords: Lung cancer screening; Early detection; Lung cancer; Low-dose CT; High-risk population
MeSH Terms: conditions — Lung Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening: Current smokers (>20 pack-years) or have quit within the past 15 years, non-smokers exposed to wood smoke more than 100 hours/year, or participants diagnosed with Chronic Obstructive Pulmonary Disease (COPD).
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Annual LDCT, lung function test (spirometry), anxiety/depression assessments, and serum biomarkers tests over 3 years. Follow-up will continue for 5 and 10 years or until event completion (cancer diagnosis, end of follow-up, or death).

SUMMARY:
This prospective study aims to detect early-stage lung cancer using low-dose computed tomography (LDCT) in Mexicans aged 50 or older who are current or former heavy smokers, non-smokers exposed to significant wood smoke, or diagnosed with COPD. Annual LDCT, spirometry, and serum biomarker tests will be conducted over 3 years, and a follow-up lasting up to 10 years.

DETAILED DESCRIPTION:
This prospective cohort study aims to detect lung cancer in early stages using LDCT scans in Mexican individuals aged 50 years or older. Eligible participants comprise current smokers with a history of ≥ 20 pack-years, former smokers who have quit within the past 15 years, non-smokers exposed to wood smoke more than 100 hours/year, or patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD).

Secondary objectives include assessing the 10-year mortality rate, the association of lung cancer with immunologic biomarkers, the demographic characterization of participants, the psychological impact of an LC screening program, the histological profiling of positive cases, lung function changes in at-risk individuals, and the clinical staging distribution at diagnosis.

The study will conduct annual LDCT scans, lung function tests (spirometry), anxiety and depression assessments, and serum biomarkers tests over 3 years. Positive LDCT results will adhere to LUNG-RADS guidelines and be managed by a multidisciplinary team. Prevention strategies, including tobacco cessation treatments, will be provided. Follow-up will continue for 5 and 10 years or until an event of completion occurs (cancer diagnosis, end of follow-up, or death).

ELIGIBILITY:
Inclusion Criteria:

Eligible participants over fifty years old and one of the next criteria:

* Current smokers (>20 pack-years)
* Former smokers (>20 pack-years) who have quit within the past 15 years,
* Non-smokers exposed to wood smoke more than 100 hours/year
* Patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD).

Exclusion Criteria:

* Subjects who cannot be examined by tomography due to physical limitations such as weight.
* History of any type of cancer within the last five years, except non-melanoma skin cancer.
* Symptoms consistent with some malignant neoplasm.
* People with a poor physical-emotional condition that reduces their life expectancy or does not ensure adherence to the study.

Elimination Criteria

• Withdrawal of informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mexican population aged over 50 years with lung cancer risk factors
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2027-03-24 (Estimated)

PRIMARY OUTCOMES:
Lung cancer incidence in Mexican population | Annually over 3-year from inclusion
  Assess the number of lung cancer detections after each round of screening.

SECONDARY OUTCOMES:
Lung cancer survival | 10-year follow-up or death from lung cancer
  Assess lung cancer mortality in participants included in the screening protocol and outside the protocol.
All-cause mortality | 10-year follow-up or death from lung cancer
  Asses all-cause mortality related to risk factors at the 3-years of LDCT screening and follow-up

OTHER OUTCOMES:
Lung cancer clinical stage | Annually over 3-year from inclusion
  Assess stage of the disease in patients detected by LDCT screening program
Serum immunological biomarkers | Annually over 3-year from inclusion
  Assess Inflammatory cytokines
Nodule detection rate | Annually over 3-year from inclusion
  Assess nodule detection rate, characteristics and outcomes detected at the screening protocol.
Chronic Obstructive Pulmonary disease (COPD) incidence rate | Annually over 3-year from inclusion
  Detect participants with a positive spirometry test that covers COPD diagnosis
Anxiety/Depression rate | Annually over 3-year from inclusion
  Asses psychological diagnosis (anxiety/depression) related to a lung cancer screening program.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta, M.D., M.Sc., Principal Investigator — Instituto Nacional de Cancerologia (INCan) Mexico
Locations (1):
- Instituto Nacional de Cancerologia (INCan) Mexico, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergman B, Aaronson NK, Ahmedzai S, Kaasa S, Sullivan M. The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30) for use in lung cancer clinical trials. EORTC Study Group on Quality of Life. Eur J Cancer. 1994;30A(5):635-42. doi: 10.1016/0959-8049(94)90535-5. PMID 8080679
- [Background] Arroyo-Hernandez M, Maldonado F, Lozano-Ruiz F, Munoz-Montano W, Nunez-Baez M, Arrieta O. Radiation-induced lung injury: current evidence. BMC Pulm Med. 2021 Jan 6;21(1):9. doi: 10.1186/s12890-020-01376-4. PMID 33407290
- [Background] Arroyo-Hernandez M, Alva-Lopez LF, Rendon A, Barroso-Villafuerte FR, Baez-Saldana R, Corona-Cruz JF, Farfan-Salazar G, Guerrero-Ixtlahuac J, Castillo-Gonzalez P, Salmon-Demongin A, Zaldivar-Crosby G, Bolano-Guerra LM, Zavala-Cruz GG, Sanchez-Gutierrez A, Rendon-Ramirez EJ, Magdaleno-Maldonado GE, Olivares-Torres CA, Lopez-Saucedo RA, Lizardo-Rodriguez AE, Ortiz-Vazquez S, Vazquez-Garcia J, Montes-Narvaez G, Pacheco-Juarez M, Arrieta-Rodriguez OG. Guia de Practica Clinica para el diagnostico temprano y la referencia oportuna del cancer de pulmon. Salud Publica Mex. 2022 Aug 26;64(5, sept-oct):530-538. doi: 10.21149/13919. Spanish. PMID 36130340
- [Background] Arroyo-Hernandez M, Zinser-Sierra JW, Vazquez-Garcia JC. [Lung-cancer screening program in Mexico]. Salud Publica Mex. 2019 May-Jun;61(3):347-351. doi: 10.21149/10326. Spanish. PMID 31276351
- [Background] Arrieta O, Arroyo-Hernandez M, Soberanis-Pina PD, Viola L, Del Re M, Russo A, de Miguel-Perez D, Cardona AF, Rolfo C. Facing an un-met need in lung cancer screening: The never smokers. Crit Rev Oncol Hematol. 2024 Oct;202:104436. doi: 10.1016/j.critrevonc.2024.104436. Epub 2024 Jul 6. PMID 38977146